CLINICAL TRIAL: NCT03129360
Title: A Randomized, Double-blind, Placebo-controlled Trial Investigating the Effects of Levetiracetam in Early Psychosis
Brief Title: Levetiracetam in Early Psychosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17-00266
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Psychosis; Schizophrenia; Schizo Affective Disorder; Schizophreniform
Keywords: Early Psychosis; Levetiracetam
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Levetiracetam 185 mg (Experimental): A single dose of 185mg of levetiracetam administered orally to participants. Participants undergo a 15-minute MRI scan using arterial spin labeling (ASL) before dosing and two hours post-dosing.
  Interventions: Drug: Levetiracetam
- Levetiracetam 500mg (Experimental): A single dose of 500mg of levetiracetam administered orally to participants. Participants undergo a 15-minute MRI scan using arterial spin labeling (ASL) before dosing and two hours post-dosing.
  Interventions: Drug: Levetiracetam
- Placebo (Placebo Comparator): A single dose of placebo administered orally to participants. Participants undergo a 15-minute MRI scan using arterial spin labeling (ASL) before dosing and two hours post-dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam is an atypical anticonvulsant that is frequently used in children and adults due to its superior tolerability, ease of use and excellent safety profile.
  Other Names: Keppra
  Arms: Levetiracetam 185 mg; Levetiracetam 500mg
Drug: Placebo — Prepared in capsules to appear identical to levetiracetam.
  Arms: Placebo

SUMMARY:
In order to establish target engagement and identify an effective dose the investigators will conduct a placebo-controlled single-dose parallel group trial of levetiracetam 185 mg and 500 mg in 24 medication-naïve early psychosis (EP) patients, measuring hippocampal activity by pulsed arterial spin labelling (ASL) pre-dose and 2 hours post-dose. The lower dose is calculated to achieve blood levels within the range that were associated with reduced hippocampal activity and improved cognition in patients with mild cognitive impairment; the higher dose is a typical antiepileptic dose. Successful demonstration of target engagement will be defined by an effect size of 0.5 or greater compared to placebo in reduction by levetiracetam of hippocampal blood flow measured by ASL. The optimal dose will be defined by maximal reduction of hippocampal perfusion in the absence of clinically-significant adverse effects. The investigators will also study 8 healthy control subjects to verify that baseline hippocampal blood flow is elevated in the sample of EP subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 16 to 35 years of age, inclusive, at time of informed consent
2. Must have experienced a first episode of non-affective psychosis within 5 years and exhibit current psychosis, as defined by a score of ≥ 2 on one of the following psychosis items on the BPRS: conceptual disorganization, suspiciousness, hallucinations, unusual thought content, or grandiosity, for at least 4 days per week for at least 4 weeks
3. Must have a diagnosis of either schizophrenia, schizoaffective disorder or schizophreniform disorder as established by a Structured Clinical Interview for DSMIV TR (SCID)
4. Must not have taken an oral antipsychotic medication within the past 4 weeks prior to study enrollment or received a long acting injectable antipsychotic within 3 times the dosing interval
5. If female and of childbearing potential, patients must:

   1. Have a negative urine pregnancy test (all females regardless of childbearing potential will be required to submit a pregnancy test)
   2. Not be nursing or planning a pregnancy for the duration of the study through 30 days after the last dosing visit
   3. Be abstinent or willing to use a reliable method of birth control from the screening visit and continue with the same method until termination from the study

Exclusion Criteria:

1. Current substance abuse or dependence for substances other than nicotine and THC (i.e., alcohol, amphetamines, barbiturates)

   1. A positive urine toxic screen (excluding THC, tricyclic antidepressants, or benzodiazepines (if prescribed))
   2. Moderate or severe cannabis use disorder
   3. Use of marijuana within the 72 hours prior to MRI scanning by self report
2. Diagnosis of major mood disorder or other Axis I disorder other than Schizophrenia, Schizoaffective Disorder or Schizophreniform Disorder
3. Current suicidal ideation. Suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the suicidal ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the Principal Investigator and/or PhD or MD level clinician completing screening visit
4. Pregnant, nursing or positive urine pregnancy test
5. Significant medical or neurological illness by history or physical exam including seizure disorder, history of loss of consciousness related to head trauma or developmental disorder including mental retardation
6. Metal implants, pacemaker, or other metal in the body or medicinal patch
7. History of claustrophobia
8. Currently taking any antipsychotic medication (within 4 weeks)

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: donald.goff@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to donald.goff@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levetiracetam 185 mg | Levetiracetam 500mg | Placebo
Started | 9 | 8 | 8
Completed | 8 | 6 | 7
Not Completed | 1 | 2 | 1
Not completed — Did not meet entry criteria | 0 | 2 | 1
Not completed — Excluded due to motion in scanner | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levetiracetam 185 mg | Levetiracetam 500mg | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.13 (5.94) | 25.17 (4.07) | 25.17 (2.35) | 25.16 (4.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 8 | 5 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6
  Not Hispanic or Latino | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 2 | 3 | 4 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Cerebral Blood Flow (CBF)
Description: CBF will be measured by Arterial Spin Labeling (ASL)
Time Frame: Baseline, 2 Hours Post-Treatment
Measure: Mean (Standard Deviation); unit: mL / (100g * min)
Arm/Group | Levetiracetam 185 mg | Levetiracetam 500mg | Placebo
Number analyzed (Participants) | 8 | 6 | 7
mL / (100g * min) | -2.21 (3.2) | -3.83 (2.29) | -1.29 (1.66)

ADVERSE EVENTS:
Time Frame: 3 Years
Description: Systematic assessment via administration of the Systematic Assessment for Treatment Emergent Side Effects (SAFTEE) questionnaire and follow-up phone call monitoring.
Arm/Group | Levetiracetam 185 mg | Levetiracetam 500mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/9 | 4/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levetiracetam 185 mg (N=9) | Levetiracetam 500mg (N=8) | Placebo (N=8)
Memory Problems (Nervous system disorders) | 0 | 1 | 0
Sedation/Drowsiness (Nervous system disorders) | 1 | 1 | 0
Hallucinations (Nervous system disorders) | 0 | 0 | 1
Dizziness (General disorders) | 0 | 1 | 0
Yelling/anger (Nervous system disorders) | 0 | 1 | 0
Night sweats/vivid dreams/overheated feeling (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03129360/Prot_SAP_000.pdf